CLINICAL TRIAL: NCT01312584
Title: The Effect of Alkalisation on the Absorption, Metabolism and Vascular Reactivity of Cocoa Flavanols
Brief Title: The Effects of Alkalised Cocoa on Human Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Dr Jeremy P E Spencer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UReading-2010-01
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2010-11

CONDITIONS: Cardiovascular Disease
Keywords: Flavanol; Cocoa; Vascular function; Absorption; Metabolism; Alkalisation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Non alkalised High Flavanol (Placebo Comparator): Non-alkalised high flavanol cocoa drink containing 1745 mg of total flavanols
  Interventions: Dietary Supplement: Processed High-flavanol
- Alkalised high Flavanol (Active Comparator): Alkalised high flavanol cocoa drink (medium alkalisation) containing 410 mg of total flavanols
  Interventions: Dietary Supplement: Processed High-flavanol
- Alkalised Low Flavanol (Active Comparator): Alkalised low flavanol cocoa drink (heavily alkalised) containing 1.26 mg of total flavanols
  Interventions: Dietary Supplement: Processed High-flavanol

INTERVENTIONS:
Dietary Supplement: Processed High-flavanol

SUMMARY:
The primary propose of this study is to determine how processing, in particular alkalisation, alters the vascular effects of high-flavanols foods such as cocoa

DETAILED DESCRIPTION:
A randomised, triple blind, cross-over design human intervention studies will be conducted in 10 healthy human volunteers to test the impact of alkalisation on the absorption, metabolism and vascular reactivity of cocoa flavanols. Participants will be requested to consume a standardised high flavanol-rich cocoa, non-alkalised (1745 mg of flavanols), a low-flavanol cocoa, heavily alkalised (1.3 mg of flavanols) and a flavanol-rich cocoa, medium alkalisation (410 mg of flavanols). The three intervention diets are otherwise matched for macro- and micronutrient content. Vascular measurements will be performed by using Flow Mediated Dilation (FMD), Laser Doppler imaging (LDI) and Digital Volume Pulse (DVP). Blood and urine samples will be taken to measure the concentration of flavonoids from the cocoa drinks and markers of blood vessel function. A number of other biochemical and physiological measures will be recorded including blood glucose, lipoproteins, cytokine levels and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male
* signed consent form
* age of 18-35 years inclusive
* BMI between 18.5-30

Exclusion Criteria:

* Blood pressure > 150/90 mmHg
* Haemoglobin (anaemia marker) < 125 g/l
* Gamma GT (liver enzymes) > 80 IU/l
* Cholesterol > 6.5 mmol/l
* Had suffered a myocardial infarction or stroke in the previous 12 months
* Suffers from any reproductive disorder
* Suffers from any blood-clotting disorder
* Suffers from any metabolic disorders (e.g. diabetes or any other endocrine or liver diseases)
* Any dietary restrictions or on a weight reducing diet
* Drinking more than 21 units per week
* On any lipid-modifying medication
* On any blood pressure lowering medication
* On any medication affecting blood clotting
* Planning on altering consumption of vitamin supplements/fish oil capsules during the course of the study
* Regular or vigorous exercise (3 times/week, 20 minutes each session)
* Smoking

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
In vivo circulatory effects relative to a non-alkalised high-flavanol cocoa. | change in Flow Mediated Dilation response between baseline and 2h
  Flow Mediated Dilation

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom